CLINICAL TRIAL: NCT02256397
Title: Home-Centered Comprehensive Care (HCCC) for Children With Severe Asthma: A Pilot Trial
Brief Title: Home Centered Comprehensive Care (HCCC) for Children With Asthma
Acronym: HCCC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Ricardo A. Mosquera, Assistant Professor of Pediatrics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HSC-MS-14-0380; UL1TR000371 (NIH); KL2TR000370 (NIH)
Record Dates: First submitted 2014-09-30; First posted 2014-10-03 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Standard comprehensive care (Active Comparator): Standard comprehensive care at High Risk Children's Clinic
  Interventions: Other: Standard comprehensive care
- Enhanced comprehensive care (Experimental): standard comprehensive care at the High Risk Children's Clinic enhaced with new technologies:
  * If between 2 and 5 years old--> will receive Home-centered comprehensive care with the propeller
  * 5 and above--> will receive home-centered comprehensive care with propeller and PIKO
  Interventions: Other: Standard comprehensive care; Other: enhanced comprehensive care

INTERVENTIONS:
Other: Standard comprehensive care — Standard comprehensive care at High Risk Children's Clinic
Other: enhanced comprehensive care — standard comprehensive care at the High Risk Children's Clinic enhaced with new technologies:
  * If between 2 and 5 years old--> will receive Home-centered comprehensive care with the propeller
  * 5 and above--> will receive home-centered comprehensive care with propeller and PIKO
  Arms: Enhanced comprehensive care

SUMMARY:
The purpose of this study is to assess whether comprehensive care enhanced with new technology to optimize asthma care in the home (using both a special sensor to track inhaler use and a hand-held PIKO-1 device to assess patients' forced expiratory volume in the 1st second [FEV1]) is effective in reducing total days when medical treatment is given outside the home (in clinic, emergency department, or hospital) among children with severe asthma receiving comprehensive care.

DETAILED DESCRIPTION:
BACKGROUND INFORMATION

Asthma is the most common pediatric chronic disease. Despite the understanding of its pathophysiology and the availability of effective therapies, adverse effects on health, school attendance, academic achievement, and family life remain high, particularly among children with severe asthma in minority or low income families.

Innovative new approaches are needed. One innovation that have shown to be cost-effective in high-risk chronically ill children, including children with severe asthma, is care in an enhanced medical home, our High-Risk Comprehensive Care (HRCC) which was designed to optimize care in medical settings. The innovation to be pilot-tested in the proposed research is Home-Centered Comprehensive Care (HCCC) designed to also optimize care in the home and thereby reduce clinic visits and school absences and further decrease Emergency Department visits and hospital days. The proposed HCCC trial builds on the infrastructure, cell phone access to the child's primary caregivers at any hour, and improved outcomes established in our previous HRCC trial (clinicaltrials.gov Identifier: NCT02128776.

DESIGN

Pilot trial of 80 children (2-18 years of age) with uncontrolled severe asthma randomized to either:

* High-Risk Comprehensive Care (HRCC) that includes 24/7 cell phone access to skilled caregivers, same day care for acute illness Monday through Friday, subspecialty care available in the same facility, and identification each weekday of all children having ED visits and hospitalizations to assure prompt follow-up and coordination of care; or
* Home-Centered Comprehensive Care (HCCC) that will also include: 1) monitoring and augmenting treatment adherence using a special sensor to track inhaler use and identify inadequate or excessive medication; 2) using a simple hand-held PIKO-1 device to assess and transmit to caregivers the 1-second forced expiratory volume, allowing caregivers to better assist the parents and to make better treatment decisions and gauge response at any hour.

HYPOTHESES

HCCC will be associated with:

1. A >40% reduction in treatment days outside the home (in a clinic, ED visits or hospital) per child-year from enrollment to the end of the trial (primary hypothesis);
2. A decrease in school absences with respiratory problems to <5 d per school year;
3. An increase in FEV1>12% in routine pulmonary function tests in our clinic at 12 mo. after enrollment;
4. Increased maternal satisfaction on the Consumer Assessment of Healthcare Providers and Systems Survey;
5. Reduced or low net health system costs relative to that reported for common treatment methods for asthma (expressed as health system cost per clinic visit, ED visit, hospitalization, or school absence prevented);
6. Reduced Medicaid costs (due to lower reimbursements for clinic, ED, and hospital care);
7. An increase in medical school costs relative to reimbursements that will be lower than the savings to Medicaid (due to its reduction in reimbursements). Such a difference will be important in efforts to promote adequate reimbursements for such care to the medical school

OBJECTIVES:

1.To randomize 80 eligible children to either standard HRCC or to HCCC in addition to HRCC in a pilot trial and evaluate whether the augmentation of the HCCC program will:

1. reduce total days when medical treatment is given outside the home (in a clinic, ED, or hospital);
2. reduce days of school missed with respiratory illnesses (including respiratory infections with symptoms aggravated by asthma);
3. improve routine pulmonary function tests one year after enrollment;
4. augment maternal satisfaction of care above even the high current levels for CC;
5. reduce costs from a health system perspective and government (Medicaid) perspective
6. increase costs relative to reimbursements from the provider (medical school) perspective

STUDY DESIGN:

Pilot trial of 80 severe asthmatics attending the HRCC that includes 24/7 cell phone access to skilled primary caregivers or to HRCC with the addition of HCCC that will also include: 1) monitoring and augmenting treatment adherence using a special sensor to track inhaler use and identify inadequate or excessive medication; 2) using a simple hand-held PIKO-1 device to assess and transmit to caregivers the 1-second forced expiratory volume, allowing caregivers to better assist the parents and to make better treatment decisions and gauge response at any hour.

The pilot trial will have duration of 2 years. We will measure efficacy based on increase FEV1 in routine pulmonary function test, reduced total days spent in clinics, Emergency departments and hospital, and well as reduced total days of school missed due to pulmonary illness. Safety will be assessed by looking at any unexpected adverse events.

With parental consent, we can also augment our care through use of Linked In to visualize the child and assess his/her condition. We recently surveyed our asthma patients given CC and to our surprise found that 75% (30/42) have access to "Linked in" on their home computer or smart phone.

ELIGIBILITY:
Inclusion Criteria:

* Children with severe asthma (poorly controlled by NIH guidelines ) who meet the inclusion criteria for HRCC (>3 ED visits, >2 hospitalizations, or >1 pediatric ICU admission in past as well as a >50% estimated risk of hospitalization in next yr).

Exclusion Criteria:

* other major lung disease (e.g. cystic fibrosis or bronchopulmonary dysplasia) or neuromuscular impairment.

Ages: 2 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 63 (Actual)
Dates: Start 2014-10; Primary Completion 2016-12 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Medical treatment outside of home | 2 years
  Total number of days when medical treatment was given outside the home (in a clinic, ED, or hospital).
  Measured by parent report every 3 months for both groups.

SECONDARY OUTCOMES:
Days of missed school | 2 years
  Total number of days of school missed with respiratory illnesses (including respiratory infections with symptoms aggravated by asthma).
  Measured by parental report on questionnaires given every 3 months
Pulmonary Function Tests. (PFTs) | 2 years
  Improve routine pulmonary function tests one year after enrollment by measuring PFTs during every clinic visit (for both groups), and by hand-held PFT device (PiKo-only for intervention group)
Parental Satisfaction | 2 years
  Parental satisfaction among groups using CAHPS survey annually.
Total costs of clinic and hospital care | 2 years
  Total cost of clinic and hospital cost measured using billing information.
Physician Services Cost to Reimbursement | 2 years
  Physician Services cost to reimbursement measured using UT claims data.

CONTACTS AND LOCATIONS:
Overall Officials: Ricardo A Mosquera, MD, Principal Investigator — University of Texas Medical School in Houston
Locations (1):
- High Risk Children's Clinic, Houston, Texas, United States